CLINICAL TRIAL: NCT00242450
Title: The Effect of Metoclopramide on Feeding in Very Low Birthweight Newborns : a Randomized, Double Blind, Placebo Controlled Pilot Study and a Proposal for a Multicentre Trial
Brief Title: Metoclopramide Use in Very Low Birth Weight Newborns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R-02-012
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2005-05

CONDITIONS: Infant, Premature
Keywords: metoclopramide; feeding; very low birthweightnewborn
MeSH Terms: conditions — Premature Birth | interventions — Metoclopramide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Metoclopramide

SUMMARY:
During the first 7 days of life very small babies will receive the drug metoclopramide or a salt solution through an intravenous line. They will also begin to receive a very small amount of breast milk or formula within the first 72 hours of life, in addition toother nourishment that is provided by an intravenous line, according to standard hospital procedure. We think that the babies who receive the medication may reach full oral feeds than babies who receive the salt solution.

DETAILED DESCRIPTION:
Clinically stable, premature babies (birth weight between 500 and 1,250g) will be randomized to receive metoclopramide (0.1 mg/kg IV q8h)or an equal volume of placebo for 7 days.A transition feeding schedule will begin within the first 72 hours of life. The time to full feeds for the 2 groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* birth weight 500 to 1,250g
* clinically stable
* no contraindications to initiating minimal enteral feeding

Exclusion Criteria:

* birth weight > 1,250g
* clinically unstable
* any major congenital anomaly
* significant GI pathology
* severe IUGR
* cholestasis

Ages: 72 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 2002-03 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Days required to attainment of full feeds.

SECONDARY OUTCOMES:
Weight at full enteral feeds (g).
Weight at discharge (g).
Duration of TPN (days).
Length of stay(days).

CONTACTS AND LOCATIONS:
Overall Officials: Orlando daSilva, MD, Principal Investigator — University of Westen Ontario
Locations (1):
- St Joseph's Hospital, London, Ontario, Canada

REFERENCES:
- [Background] Kearns GL, van den Anker JN, Reed MD, Blumer JL. Pharmacokinetics of metoclopramide in neonates. J Clin Pharmacol. 1998 Feb;38(2):122-8. doi: 10.1002/j.1552-4604.1998.tb04400.x. PMID 9549642